CLINICAL TRIAL: NCT02311010
Title: Influence of Recipient Cytochrome P450 3A5 Polymorphism on the Metabolism of Prolonged Release Tacrolimus Administered de Novo After Renal Transplantation
Brief Title: Practical Use of Advagraf de Novo After Kidney Transplantation According to Recipient Genetic Polymorphism
Acronym: CYRANO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Prof Martine De Meyer, MD, Université Catholique de Louvain
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BE-02-RG-234; 2011-004276-11 (EudraCT Number)
Record Dates: First submitted 2014-08-21; First posted 2014-12-08 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Kidney Diseases
Keywords: transplant; immunosuppressive drug
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CYP 3 A 5 *3/*3 control group (No Intervention): CYP 3 A 5 *3/*3 control group will receive 0,20 mg/kg of Advagraf®
- CYP 3 A 5 *3/*3 (Active Comparator): CYP 3 A 5 *3/*3 will receive 0,25 mg/kg of Advagraf®
  Interventions: Drug: Advagraf
- CYP 3 A 5 *1/*3 (Active Comparator): CYP 3 A 5 *1/*3 will receive 0,30 mg/kg of Advagraf®
  Interventions: Drug: Advagraf
- CYP 3 A 5 *1/*1 (Active Comparator): CYP 3 A 5 *1/*1 will receive 0,35 mg/kg of Advagraf®
  Interventions: Drug: Advagraf

INTERVENTIONS:
Drug: Advagraf — daily dose adapted according to Cyp 3A5 polymorphism
  Other Names: Tacrolimus prolonged release formulation
  Arms: CYP 3 A 5 *1/*1; CYP 3 A 5 *1/*3; CYP 3 A 5 *3/*3

SUMMARY:
To optimize the Advagraf (tacrolimus once a day) initial daily dose used in de novo after kidney transplantation in combination with MMF (or MPA) and corticosteroids (CS) regarding of the genetic Cyp 450 3A5 polymorphism of the recipient.

The study of the tacrolimus through level (ng/ml) determines if the therapeutic level is reached.

ELIGIBILITY:
Inclusion Criteria:

* First or second Kidney Transplantation from deceased or living donor

Exclusion Criteria:

* Donor age < 5 years.
* Patients who require plasma exchange because of high immunological risk

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics of tacrolimus | 1 year
  tacrolimus level (ng/ml) at C0 every 3 days during 2 weeks and thereafter every month during 1 year

SECONDARY OUTCOMES:
Kidney graft function | 1 year
  serum creatinine level (mg/dl) and GFR (ml/min)

OTHER OUTCOMES:
Administration strategy | first day
  starting tacrolimus daily dose (mg/kg/d) accorded to CYP 3A5 polymorphism of the recipient
New onset of diabetes after transplantation (NODAT) | 1 year
  fasting glycemia (mg/dl) HbA1C (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint Luc Université Catholique de Louvain, Brussels, Belgium

REFERENCES:
- [Derived] De Meyer M, Haufroid V, Kanaan N, Darius T, Buemi A, De Pauw L, Eddour DC, Wallemacq P, Mourad M. Pharmacogenetic-based strategy using de novo tacrolimus once daily after kidney transplantation: prospective pilot study. Pharmacogenomics. 2016 Jun;17(9):1019-27. doi: 10.2217/pgs-2016-0005. Epub 2016 Jun 8. PMID 27266721